CLINICAL TRIAL: NCT07207941
Title: Effect of Probiotics on Quality of Life, Activities of Daily Living and Anxiety in Post Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: B-Crobes Laboratory Sdn. Bhd (Unknown)
Responsible Party: Principal Investigator, Tan Hui Jan, Consultant Neurologist, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JEP-2025-671
Record Dates: First submitted 2025-09-16; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: stroke; probiotic; quality of life; anxiety; activities of daily living
MeSH Terms: conditions — Stroke; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Intervention group HEXBIO MCP Granule probiotics (Lactobacillus acidophilus, L. casei, L. lactis, Bifidobacterium bifidum, B. infantis, B. longum), one sachet twice daily for 3 months.
  Interventions: Dietary Supplement: Hexbio
- Placebo (Placebo Comparator): Placebo Control Matching placebo sachets, identical in appearance and schedule.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Hexbio — HEXBIO MCP Granule probiotics (Lactobacillus acidophilus, L. casei, L. lactis, Bifidobacterium bifidum, B. infantis, B. longum), one sachet twice daily for 3 months.
  Arms: Intervention
Other: Placebo — Matching placebo sachets, identical in appearance and schedule
  Arms: Placebo

SUMMARY:
Research on Effect of probiotics on quality of life, activities of daily living and anxiety in post stroke patients

DETAILED DESCRIPTION:
Background:

Stroke survivors often experience reduced quality of life (QoL), impaired activities of daily living (ADL), and high levels of anxiety. Emerging evidence suggests that modulation of the gut-brain axis through probiotics may improve neuropsychological and functional outcomes. However, data from Malaysian populations are lacking.

Objective:

To evaluate the effects of probiotic supplementation compared to placebo on QoL, ADL, anxiety symptoms, and functional outcomes in post-stroke patients.

Study Design:

This is a single-center, randomized, double-blind, placebo-controlled clinical trial.

Methods:

A total of 110 patients with moderate ischemic stroke (mRS 2-4) within 3 months of onset will be recruited from the Neurology Clinic, Hospital Canselor Tuanku Muhriz, Kuala Lumpur. Participants will be randomized (1:1) to receive either:

* Intervention: HEXBIO MCP Granule probiotics (Lactobacillus acidophilus, L. casei, L. lactis, Bifidobacterium bifidum, B. infantis, B. longum), one sachet twice daily for 3 months.
* Control: Matching placebo sachets, identical in appearance and schedule. Both groups will continue standard stroke treatment. Primary outcome is QoL measured using the Stroke-Specific Quality of Life (SS-QoL) scale. Secondary outcomes include ADL (Barthel Index), anxiety symptoms (GAD-7), and functional status (mRS score). Assessments will be performed at baseline and 3 months.

Sample Size:

A total of 110 patients (55 per arm) will provide sufficient power to detect clinically meaningful differences, accounting for a 5% dropout rate.

Data Analysis:

Intention-to-treat analysis will be conducted using SPSS v26. Between-group differences will be assessed using appropriate parametric or non-parametric tests, with significance set at p < 0.05.

Study Duration:

Recruitment will begin in Sept 2025 and is expected to complete by May 2028.

Expected Impact:

This study will provide new evidence on the role of probiotics in improving QoL, daily functioning, and psychological well-being among Malaysian post-stroke patients, potentially informing adjunctive rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with moderate ischemic stroke with mRS score of 2-4 from onset of stroke up to 3 months.
* Patients aged 18 to 80 years, who are able to read and write in English and/or Bahasa Malaysia
* Provide informed consent

Exclusion Criteria:

* Patients with aphasia
* Patients who have received thrombolysis or mechanical thrombectomy
* Gastrointestinal related diseases such as lactose intolerance, coeliac disease, Renal or hepatic insufficiency (Based on recent six-month blood profile)
* Progressive neurological disease (Alzheimer's disease, Parkinson's Disease, Motor Neuron Disease)
* Pregnancy and breastfeeding.
* Secondary cause of stroke- vasculitis, cerebral venous sinus thrombosis, connective tissue disorders
* Past history of psychiatric disorders (depression, anxiety)
* Recent use of probiotics and allergies to probiotics
* Immunosuppressed patients (HIV, malignancy)
* Patient with septicemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 3 months
  QoL measured using the Stroke-Specific Quality of Life (SS-QoL) scale. To assess the patient's quality of life, validated Stroke Specific Quality of life (SS-QoL) questionnaire in English version will be used. This questionnaire consists of 12 domains which includes energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision, and work/productivity. Each question is scored using 5 point Likert scale and the total score is calculated which can range from 49-245. The higher the score, better the quality of life. This questionnaire is validated and requested for permission.

SECONDARY OUTCOMES:
Secondary objectives: Activities of daily living | 3 months
  Activities of daily living is measured using Barthel Index (BI) which contains of 10 items. BI is a measurement scale used to assess an individual's ability to perform activities of daily living (ADL) and mobility. The score ranges from 0-10 and the overall score is calculated. The higher the score, better the functional status.
Secondary objective: Anxiety Score | 3 months
  Anxiety score is calculated using Generalised Anxiety Disorder- 7 (GAD-7) score. GAD 7 is a screening tool and it has 7 items with score ranging from 0-3 for each item and the total score is calculated. The higher the score, the worse the anxiety symptoms. A score of 10 indicates anxiety.
Secondary objective: modified Rankin scale | 3 months
  Modified Rankin Scale (mRS) assess functional recovery and independence after stroke. It uses a 5 point scale, where a higher scale indicates more severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Nasir Shafiee, Study Director — National University of Malaysia
Locations (1):
- National University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Study has not commenced